CLINICAL TRIAL: NCT06050525
Title: Incidence of Acute Kidney Injury and Risk Factors in Newborns With Congenital Diaphragmatic Hernia
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Urban Fläring, M.D. Ph.D. Associate Professor., Karolinska Institutet
Other Study IDs: K 2023-7065
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Congenital Diaphragmatic Hernia; Acute Kidney Injury; Multiple Organ Failure; Pulmonary Hypertension; Hyperchloremia
Keywords: Congenital Diaphragmatic Hernia; Acute Kidney Injury
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Acute Kidney Injury; Multiple Organ Failure; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this project is to elucidate the incidence of acute kidney injury (AKI) in newborns with congenital diaphragmatic hernia during stay in the Pediatric intensive care unit. (PICU). This patient group often presents with severe circulatory and respiratory dysfunction requiring intensive care treatment. Characterization of risk factors to AKI will also be performed.

DETAILED DESCRIPTION:
There is an overwhelming number of studies showing that complication with acute kidney injury (AKI) in critically ill patients, including children and newborns results in increased morbidity and mortality. The more severe AKI, the higher risk of bad outcome. In the neonatal intensive care unit (NICU), the incidence of AKI is approximately 30 %, even higher in full-term babies (36 %).

Newborns with congenital diaphragmatic hernia (CDH) often present with severe cardio-respiratory dysfunction, often complicated by pulmonary hypertension (PPHN) requiring mechanical ventilation and vasoactive/inotropic drugs, especially during the first week in the intensive care. Some of these patients deteriorates and cannot maintain vital parameters despite conventional treatment and will therefore require extra corporeal membrane oxygenation). During the ICU-stay, the patients are subjected to several risk factors for developing AKI. Among physiological risk factors, PPHN, low oxygenation and blood pressure may result in renal dysfunction. Iatrogenic factors include the need for nephrotoxic drugs, not least antibiotics (Vancomycin, Gentamycin) and antimycotics. In addition, hyperchloremia may contribute to the development of AKI, since impaired renal blood flow is associated with hyperchloremia. The AKI incidence and its risk factors in CDH patients is not well studied.

The objectives of this well characterized retrospective cohort study is to establish AKI incidence in critically ill CDH-patients and investigate possible associations between risk factors and AKI (exposure to nephrotoxic drugs, degree of multiple organ failure, PPHN, vasoactive/inotropic requirement, oxygenation index, fluid overload and hyperchloremia) during PICU stay. The association of the risk factors to different stages of AKI will also be investigated.

ELIGIBILITY:
Inclusion Criteria: Newborns with congenital diaphragmatic hernia intubated and started invasive ventilation within 2 days.

-

Exclusion Criteria:

* Invasive ventilation initiated after 2 days.
* Severe comorbidity not compatible with life and/or not possible to correct surgically.
* Death occurring within 2 days.

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with congenital diaphragmatic hernia, intubated and started invasive ventilation within 2 days, referred to Karolinska University Hospital, Stockholm, Sweden.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury in newborn patients with congenital diaphragmatic hernia (CDH) (n=108) | Acute kidney injury evolving during PICU-stay (from birth up to 10 weeks, which is the longest PICU-stay among the patients).)
  Patients having or not having acute kidney injury will be determined by the score: neonatal Kidney Diseases: Improving Global Outcomes (n-KDIGO), based upon creatinine concentration (mikromoles/L). A 1.5-fold increase in creatinine concentration increase from first sampling will be classified as acute kidney injury.

SECONDARY OUTCOMES:
Pulmonary hypertension | Developing during PICU-stay (from birth up to 10 weeks)
  A patient is classified as having PPHN on the first echocardiogram if the right ventricular systolic blood pressure is 67% or more of the systemic blood pressure. Acute kidney injury will be determined using n-KDIGO described in Primary Outcome Measure. In the statistic analysis, the variables will be dichotomous. Possible association will be analysed using logistic regression analysis in this cohort of newborn patients with CDH (n=108)
Use of nephrotoxic drugs | Given during PICU-stay (from birth up to 10 weeks)
  If given 3 days or more during PICU-stay, Nephrotoxic drugs (Vancomycin, Meropenem, Gentamycin, Amphotericin B, Tazobactam and Fluconazole) will be investigated using logistic regression analysis to elucidate if there is an association with the development of acute kidney injury (defined by n-KDIGO) in this cohort of newborn patients with CDH (n=108)
Duration (days during first week in the PICU) of hyperchloremia | From birth up to one week in the. PICU.
  Plasma chloride concentration has been obtained from blood gas analysis on a daily basis during the first week in the PICU. It will be investigated if days with a chloride concentration >110mmol/L is associated with the development of acute kidney injury (defined by n-KDIGO) using logistic regressionin this cohort of newborn patients with CDH (n=108)
Development of multiple organ failure. | From birth up to one week in the PICU
  Maximum development of multiple organ failure during the first week in the PICU will be determined defined by the PEdiatric Logistic Organ Dysfunction Score (PELOD-2-score). Higher values means a worse. outcome. A possible association between PELOD-2 score and the development of acute kidney injury will be investigated using logistic regression in this cohort of newborn patients with CDH (n=108)
Mortality during PICU-stay (max 10 weeks). | PICU-stay. (up to 10 weeks).
  Association between the development of acute kidney injury defined by n-KDIGO and mortality occurring during PICU stay will be investigated using logistic regression in this cohort of newborn patients with CDH (n=108)

CONTACTS AND LOCATIONS:
Overall Officials: Urban Fläring, MD. Ph.D., Principal Investigator — Department of Pediatric Anesthesia and Intensive Care. Karolinska University Hospital. Stockholm. Sweden.
Locations (1):
- Department of Pediatric Anesthesia and Intensive Care. Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Barhight MF, Lusk J, Brinton J, Stidham T, Soranno DE, Faubel S, Goebel J, Mourani PM, Gist KM. Hyperchloremia is independently associated with mortality in critically ill children who ultimately require continuous renal replacement therapy. Pediatr Nephrol. 2018 Jun;33(6):1079-1085. doi: 10.1007/s00467-018-3898-2. Epub 2018 Feb 5. PMID 29404689
- [Result] Jetton JG, Boohaker LJ, Sethi SK, Wazir S, Rohatgi S, Soranno DE, Chishti AS, Woroniecki R, Mammen C, Swanson JR, Sridhar S, Wong CS, Kupferman JC, Griffin RL, Askenazi DJ; Neonatal Kidney Collaborative (NKC). Incidence and outcomes of neonatal acute kidney injury (AWAKEN): a multicentre, multinational, observational cohort study. Lancet Child Adolesc Health. 2017 Nov;1(3):184-194. doi: 10.1016/S2352-4642(17)30069-X. PMID 29732396
- [Result] Chatterjee D, Ing RJ, Gien J. Update on Congenital Diaphragmatic Hernia. Anesth Analg. 2020 Sep;131(3):808-821. doi: 10.1213/ANE.0000000000004324. PMID 31335403
- [Result] Liberio BM, Brinton JT, Gist KM, Soranno DE, Kirkley MJ, Gien J. Risk factors for acute kidney injury in neonates with congenital diaphragmatic hernia. J Perinatol. 2021 Aug;41(8):1901-1909. doi: 10.1038/s41372-021-01119-1. Epub 2021 Jun 12. PMID 34120147